CLINICAL TRIAL: NCT01574677
Title: Assessment of Septin9 Biomarker for Detection of Colorectal Cancer in Patients With Positive Fecal Immunochemical Test
Status: Withdrawn | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Collaborators: Kaiser Permanente (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: Septin 9 Colorectal Biomarker
Record Dates: First submitted 2012-03-20; First posted 2012-04-10 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; fecal immunochemical test; Septin 9; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Screening FIT positive: Patients aged 49-80, with a positive screening FIT, who are referred to colonoscopy, and who meet inclusion criteria.

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer death in the United States and affects men and women almost equally. The United States Preventative Services Task Force (USPSTF) currently recommends screening with any of three options, which include fecal testing, flexible sigmoidoscopy, or colonoscopy.

Screening for CRC with fecal occult blood testing (using a guaiac-based test) done annually or biennially has been shown to decrease mortality 15-33% primarily through detection of early stage cancer. Guaiac fecal occult blood testing (gFOBT) has a known positive balance of benefit and risk in screening populations, is the least expensive, and is the preferred method of screening in 30-55% of patients. The fecal immunochemical test (FIT) offers significant improvements over the gFOBT, most notably that it is easier to use (requires fewer samples and no dietary or medication restrictions) and is more sensitive than the gFOBT with respect to detecting both CRC and precancerous adenomas. As a result of improved test performance and usability, in 2008 multiple professional societies endorsed the use of four types of FITs for colorectal cancer screening. Kaiser Permanente currently uses the OC-Micro FIT as the fecal screening test in all regions.

In recent years, intensive efforts have been undertaken to identify blood-based markers that may provide a promising alternative or supplement to fecal testing for non-invasive CRC screening. One method under development is to identify aberrantly methylated genes in cancer tissue through a blood test. Prior studies have explored those specific colorectal cancer genes that show the highest differences in methylation between the cancer and background genetic expression. Of these, methylation of the Septin 9 gene through a qPCR assay is relatively well studied.

The proposed study aims to evaluate whether the Septin 9 biomarker may be used to supplement the OC-Micro FIT for colorectal cancer screening in such a way as to safely reduce unneeded colonoscopies. The population of interest for this study-those with a positive screening OC-Micro fecal immunochemical test-has a CRC prevalence of approximately 5%. Knowing how well Septin 9 can identify those without cancer prior to colonoscopy is important largely because colonoscopy, even when done diagnostically (e.g., after a positive FIT result), can cause serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 49-80
* Member of Kaiser Permanente Northwest or Southeast
* English or Spanish speaking
* Had a positive fecal screening (FIT) and has an active referral to colonoscopy

Exclusion Criteria:

* Having a personal history of colon cancer
* Having had a prior colonoscopy within 5 years
* Currently under hospice care
* Currently in a skilled nursing facility
* Currently being treated for active cancer (any type)
* Having ever had carcinoid tumor or full colectomy
* Having indicated a preference at enrollment into Kaiser health plan to not participate in research

Ages: 49 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be identified at Kaiser Permanente Northwest (KPNW) and Kaiser Permanente Georgia (KPGA). KPNW is a nonprofit group-model HMO with membership of about 485,000 in SW Washington and NW Oregon. KPNW includes 797 physician s and 395 allied clinicians (265 primary care providers). The member population base is similar to the local insured community in terms of age, gender, race, and ethnicity. About 19% of members are racial and ethnic minorities. Membership of KPGA has a racial and socioeconomic distribution similar to metropolitan Atlanta: ~ 50% Caucasian, 45% African American, 4% Hispanic, and 1% other races. 90 percent of the KPGA membership receives primary care at 12 medical offices owned and operated by KPGA and through contracts with 125 community practices.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06

PRIMARY OUTCOMES:
Performance characteristics of the Septin 9 biomarker among patients who have a positive FIT result | Participants are prospectively enrolled. Eligible participants will be asked to provide a blood sample at least 2 days prior to receiving a colonoscopy. The timeframe for participation will generally be within 3 months of receiving a positive FIT result.
  Sensitivity, specificity, positive predictive value, and negative predictive value of Septin 9 (relative to colonoscopy) for detecting CRC in a sample of individuals with a positive test result for single-sample OC-Micro FIT using various thresholds for Septin 9 positivity.

SECONDARY OUTCOMES:
Concordance and discordance (Kappa scores) between Septin 9 test results and colonoscopy findings associated with patient demographic factors. | The timeframe for participation will generally be within 3 months of receiving a positive FIT result.
  Patient demographic factor such as age and gender will be assessed.
Concordance and discordance (Kappa scores) between Septin 9 test results and colonoscopy findings associated with co-morbid conditions. | The timeframe for participation will generally be within 3 months of receiving a positive FIT result.
  Co-morbid conditions will include, for example, diabetes, congestive heart failure, etc.
Concordance and discordance (Kappa scores) between Septin 9 test results and colonoscopy findings associated with specific medication use practices. | The timeframe for participation will generally be within 3 months of receiving a positive FIT result.
  Medications will include common medications in screening population (ie. blood thinners).

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Coronado, PhD, Principal Investigator — Kaiser Permanente, Center for Health Research NW; Amanda Petrik, Study Director — Kaiser Permanente Center for Health Research NW
Locations (2):
- United States (2):
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - Kaiser Permanente Northwest, Portland, Oregon